CLINICAL TRIAL: NCT02675205
Title: Ticagrelor Versus Clopidogrel for Platelet Inhibition in Patients Undergoing Neurovascular Stenting for Intracranial Aneurysm
Brief Title: Ticagrelor vs Clopidogrel for Platelet Inhibition in Stenting for Cerebral Aneurysm
Acronym: TIC-TAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGR_2014-33; 2014-005720-10 (EudraCT Number)
Record Dates: First submitted 2015-12-30; First posted 2016-02-05 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Clopidogrel; Ticagrelor; Aspirin

ARMS (2):
- clopidogrel-aspirin (Active Comparator): clopidogrel: 75mg and aspirin 250 mg once a day for 15 weeks; prescribed 3 weeks before surgery.
  Interventions: Drug: Clopidogrel; Drug: aspirin
- ticagrelor-aspirin (Experimental): Ticagrelor: 90 mg bid and aspirin 250 mg once a day for 15 weeks; prescribed 3 weeks before surgery
  Interventions: Drug: Ticagrelor; Drug: aspirin

INTERVENTIONS:
Drug: Clopidogrel — clopidogrel: efficacy and safety in cerebral aneurysm stenting
  Arms: clopidogrel-aspirin
Drug: Ticagrelor — ticagrelor:efficacy and safety in cerebral aneurysm stenting
  Arms: ticagrelor-aspirin
Drug: aspirin

SUMMARY:
Part of interventional neuroradiology procedures for the treatment of selected cerebral aneurysms are now based on stenting. To reduce thromboembolic events, dual antiplatelet therapy (APT) combining aspirin and clopidogrel is proposed with close monitoring, since 1/3 of the patients are low responders due to variation of the biological response to clopidogrel . Ticagrelor is used by few teams but has never been evaluated in a randomized controlled trial. It could be an option for APT due to more reproducible response with less interindividual variability and reduced monitoring. The aim of this study is to demonstrate the interest of ticagrelor for the dual APT for platelet inhibition, in patients undergoing neurovascular stenting for cerebral aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* unruptured cerebral aneurysm
* elective endovascular treatment
* stenting required
* dual antiplatelet therapy required

Exclusion Criteria:

-none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
proportion of patients requiring at least one change of drug or dose adjustment to achieve platlet functional inhibition | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France